CLINICAL TRIAL: NCT03217552
Title: An Observational Study to Evaluate the Diagnostic and Predictive Accuracy of the Mologic Biomarker Panel in Patientsrnwith Severe Infection
Brief Title: The Performance of the Mologic Biomarker Panel in Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mologic Ltd (Industry)
Collaborators: University College London Hospitals (Other); Innovate UK (Other Government)
Responsible Party: Sponsor
Other Study IDs: CN010
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Sepsis; Infection
MeSH Terms: conditions — Sepsis; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- The Emergency Department: The study aims to evaluate the test in this environment as a potential diagnostic. All patients will be screened using the electronic patient management system within the ED.
  A single sample of approximately 20ml of blood, will be obtained at the same time as a clinically indicated blood culture (triggered by clinician concern for infection). The sample will be processed as described in the laboratory manual, aliquoted and frozen for future batch analysis. This analysis will include:
  * The Mologic Biomarker Panel
  * PCT
  * CRP
  * Other inflammatory markers or pathogen detection that may augment the panels accuracy
  All conventional standard of care testing will be done at the study site as part of the enrolled subject's routine clinical care.
  Interventions: Diagnostic Test: Mologic Biomarker Panel
- Critical Care Unit: Two patient populations admitted to the CCU will be approached for inclusion into the study:
  * Patients being managed for potential infection
  * Patients having undergone elective major surgery and admitted to the CCU as part of their care pathway. These patients will act as controls as the majority show signs and symptoms of inflammation but rarely develop an infection.
  Patients with potential infection: UCLH Critical Care Unit has approximately 1000 emergency admissions per year. Complicated infection (sepsis or septic shock) being the commonest underlying reason for admission.
  Interventions: Diagnostic Test: Mologic Biomarker Panel
- Patients undergoing major surgery: UCLH Critical Care admits approximately 1000 patients per year following major elective surgery. These patients frequently exhibit the features of SIRS but the incidence of infection/sepsis is low (approximately 5%) and very rare in the first 3 days' post-surgery. This group is to be studied as a negative control group to ensure the Mologic Biomarker Panel is able to detect the difference between the similar inflammatory phenotypes developed through infection and surgical trauma.
  Interventions: Diagnostic Test: Mologic Biomarker Panel

INTERVENTIONS:
Diagnostic Test: Mologic Biomarker Panel — In brief the proposed biomarkers will be measured in the laboratory of Mologic . These will initially be performed using standard lab assays (Enzyme Linked Immunosorbent Assays, ELISA). Biomarkers that show promise will then be mounted on a novel lateral flow device (under development), that could ultimately be deployed at the patients bedside.

SUMMARY:
This study is a prospective, single center, observational, cohort study of patients to determine whether the Mologic Biomarker Panel can identify patients with infection from those without, including those with other reasons for inflammation (e.g. post-operative). It will also assess whether it has the potential to judge the severity of illness, prognosticate outcome and guide antibiotic therapy.

The aim is to recruit patients who are "representative" of patients with suspected sepsis, uncomplicated infection, or non-infection related critical illness that require critical care intervention and assessment.

This study is observational and will not alter patient management or the standard of care. The results from the investigational Mologic Biomarker Panel and associated research assays will not be provided to treating clinicians, or used in any manner to affect patient care.

The study will take place over approximately an 18-month period and it is anticipated that approximately 600 patients will be collectively enrolled. The study aims to recruit patients from three environments within UCLH:

* The Emergency Department.
* Critical Care Unit
* Patients undergoing major surgery

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Investigated for potential infection (the clinical need for a blood culture)

Exclusion Criteria:

* <18 years old
* Severe anaemia (<60g/dl) and contra-indication to transfusion
* Unable to gain consent or agreement
* Treated with palliative intent
* Blood culture indicated for screening or monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe infection from:
  * The Emergency Department
  * Critical Care Unit
  * Patients undergoing major surgery
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-11-26 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Biomarkers and results from routine clinical testing for infection | 18 months
  Research assay will be used to test for the investigational Mologic biomarker panel and these results will be assessed using the results obtained from conventional testing used to identify infection (such as white cell count and CRP), in order to find a clinical association with the mologic biomarkers and patients with infections.

CONTACTS AND LOCATIONS:
Overall Officials: David Brealey, PhD MRCP FRCA, Principal Investigator — University College London Hospital
Locations (1):
- University College London Hospital, London, United Kingdom